CLINICAL TRIAL: NCT02123394
Title: Efficacy of the Mckenzie Method in Patients With Chronic Non-Specific Low Back Pain: A Randomized Placebo-Controlled Trial
Brief Title: Efficacy of the Mckenzie Method in Patients With Chronic Non-Specific Low Back Pain
Acronym: Mckenzie
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Luciola da Cunha Menezes Costa, Associate Professor, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FAPESP200755
Record Dates: First submitted 2014-04-16; First posted 2014-04-25 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Non-specific Chronic Low Back Pain
Keywords: Low Back Pain; Mechanical Low Back Pain; Low Back Ache; Low Backache; Lower Back Pain; Lumbago
MeSH Terms: conditions — Low Back Pain | interventions — Placebo Effect; Nocebo Effect

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): The patients allocated to the Placebo group will be treated with detuned pulsed ultrasound for 5 minutes and detuned short wave diathermy in pulsed mode for 25 minutes. Patients will receive 10 sessions of treatment over a period of five weeks (two sessions/week).
  Interventions: Other: Placebo
- McKenzie method (Experimental): The patients of the McKenzie group will be treated according to the principles of the method and the choice of therapeutic intervention will be guided by the physical examination findings and classification. Patients will also receive written instructions from the Treat Your Own Back book and will be asked to perform home exercises based on the principles of McKenzie method. Patients will receive 10 sessions of treatment over a period of five weeks (two sessions/week).
  Interventions: Other: McKenzie method

INTERVENTIONS:
Other: Placebo — The patients allocated to the Placebo group will be treated with detuned pulsed ultrasound therapy for 5 minutes and detuned short wave diathermy in pulsed mode for 25 minutes. Patients will receive 10 sessions of treatment over a period of five weeks (two sessions/week).
  Other Names: Placebo effect; Nocebo effect
  Arms: Placebo
Other: McKenzie method — The patients of the McKenzie group will be treated according to the principles of the method and the choice of therapeutic intervention will be guided by the physical examination findings and classification. Patients will also receive written instructions from the Treat Your Own Back book and will be asked to perform home exercises based on the principles of McKenzie method. The description of the exercises that will be prescribed in this study are already published elsewhere. Compliance with home exercises will be monitored by means of a daily-log that the patient will fill in at home and bring to the therapist at each subsequent session. Patients will receive 10 sessions of treatment over a period of five weeks (two sessions/week).
  Other Names: McKenzie
  Arms: McKenzie method

SUMMARY:
The purpose of this study is to assess the efficacy of the McKenzie method in patients with chronic non-specific low back.

DETAILED DESCRIPTION:
One hundred and forty-eight patients will be randomly allocated to two treatment groups: McKenzie method or Placebo (detuned ultrasound and short wave therapy) for 5 weeks (total of 10 sessions of 30 minutes each).

The clinical outcomes will be obtained at the completion of treatment (5 weeks) and at 3, 6, and 12 months after randomization. The data will be collected by a blinded assessor. The statistical analysis will follow the intention-to-treat principles and the between-group differences will be calculated by constructing mixed linear models.

ELIGIBILITY:
Inclusion Criteria: patients seeking care for chronic non-specific low back pain (defined as pain or discomfort between the costal margins and the inferior gluteal folds, with or without referred symptoms in the lower limbs, for at least 3 months), with a pain intensity of at least 3 points measured by a 0-10 points pain numerical rating scale, aged between 18 and 80 years and able to read in Portuguese.

-

Exclusion Criteria: patients will be excluded if they have any contraindication to physical exercise or ultrasound or short wave therapy, evidence of nerve root compromise (i.e one or more of motor, reflex or sensation deficit), serious spinal pathology (such as fracture, tumor, inflammatory and infectious diseases), serious cardiovascular and metabolic diseases, previous back surgery and pregnancy.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 5 weeks after randomization
  Pain Intensity will be measured by an 11-point (0-10) Numerical Rating Scale (Pain NRS)
Disability | Five weeks after randomization
  Disability will be measured by the 24-item Roland Morris Disability Questionnaire

SECONDARY OUTCOMES:
Pain Intensity | 3, 6 and 12 months after randomization
  Pain Intensity will be measured by an 11-point (0-10) Numerical Rating Scale (Pain NRS)
Disability | 3, 6 and 12 months after randomization
  Disability will be measured by the 24-item Roland Morris Disability Questionnaire
Function | Five weeks, 3, 6 and 12 months after randomization
  Disability and function will be measured by an 11-point (0-10) Patient-Specific Functional Scale
Kinesiophobia | Five weeks, 3, 6 and 12 months after randomization
  Kinesiophobia will be measured by the Tampa Scale of Kinesiophobia by means of 17 questions that deal with pain and intensity of symptoms.
Global perceived effect | Five weeks, 3, 6 and 12 months after randomization
  Global perceived effect will be measured by an 11-point (-5 to +5) Global Perceived Effect Scale

OTHER OUTCOMES:
Patient's expectancy for improvement | Baseline
  Will be assessed by the Expectancy of Improvement Numerical Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo OP Costa, PhD, Principal Investigator — Universidade Cidade de São Paulo; Luciola CM Costa, PhD, Study Director — Universidade Cidade de São Paulo
Locations (1):
- Universidade Cidade de Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Garcia AN, Costa LDCM, Hancock MJ, Souza FS, Gomes GVFO, Almeida MO, Costa LOP. McKenzie Method of Mechanical Diagnosis and Therapy was slightly more effective than placebo for pain, but not for disability, in patients with chronic non-specific low back pain: a randomised placebo controlled trial with short and longer term follow-up. Br J Sports Med. 2018 May;52(9):594-600. doi: 10.1136/bjsports-2016-097327. Epub 2017 Jul 12. PMID 28701365
- [Derived] Garcia AN, Costa Lda C, Hancock MJ, de Almeida MO, de Souza FS, Costa LO. Efficacy of the McKenzie method in patients with chronic nonspecific low back pain: a protocol of randomized placebo-controlled trial. Phys Ther. 2015 Feb;95(2):267-73. doi: 10.2522/ptj.20140208. Epub 2014 Oct 2. PMID 25278336